CLINICAL TRIAL: NCT03906253
Title: Effectiveness of Fractionated Laser Resurfacing to Protect Geriatric Skin From Actinic Neoplasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wright State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06438
Record Dates: First submitted 2019-04-04; First posted 2019-04-08 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Actinic Keratoses; Aging; Non-Melanoma Skin Cancer
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Factionated Laser Resurfacing - Right Arm (Experimental): Right forearm treatment of fractionated laser resurfacing.
  Interventions: Device: Fractionated Laser Resurfacing
- Factionated Laser Resurfacing - Left Arm (Experimental): Left forearm treatment of fractionated laser resurfacing.
  Interventions: Device: Fractionated Laser Resurfacing

INTERVENTIONS:
Device: Fractionated Laser Resurfacing — A rejuvenating laser that makes tiny holes in the very superficial part of the skin.

SUMMARY:
This study is following up on previous studies that have demonstrated that geriatric subjects respond different to ultraviolet B (UVB) light than young subjects. The treatment of geriatric skin with dermal rejuvenation therapies (dermabrasion, fractionated laser resurfacing) restores the appropriate UVB response. Ongoing studies have tested the ability of fractionated laser resurfacing (FLR) to assess how long this wounding effect lasts-and have found that this appears to be a durable response which lasts for at least two years. The findings that FLR protects geriatric skin at two years is the impetus for this study.

This study is an interventional study to assess if FLR treatment of one forearm of geriatric subjects with multiple actinic keratosis will result in the short-term removal of actinic keratosis, and the long-term decrease in levels of future actinic keratosis and other non-melanoma skin cancers in comparison to the untreated arm.

Study length and visit: The first part of the study is completed in 1 day then there are follow up visits at 90 days and every 6 months for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Actinic Keratosis within the past 6 months
* At least 60 years of age, or older
* Ability to comprehend procedures and risks versus benefits
* Able to provide Informed Consent
* Fair Skin (Fitzpatrick Type I or II)
* Possess both Right and Left Forearms

Exclusion Criteria:

* Uncontrolled Diabetes Mellitus
* Not able to comprehend procedures or risks versus benefits
* Pregnant or nursing
* Large tattoos on forearms
* History of abnormal healing or scarring (i.e., keloids)
* Any disease that gets worse while in the sun
* Use of topical or oral anti-inflammatory medication or steroids
* Allergy to lidocaine
* Current use of photosensitizing medication

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2018-01-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Number of Actinic Keratosis due to FLR treatment. | up to 5 years
  Investigator will assess the number of actinic keratosis on both forearms.
Change From Baseline in the Number Non-Melanoma Skin Cancers due to FLR treatment. | up to 5 years
  Investigator will assess the number of actinic keratosis on both forearms.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey B Travers, MD, PhD, Principal Investigator — Wright State University
Locations (1):
- Dayton VA Medical Center, Dayton, Ohio, United States

REFERENCES:
- [Derived] Spandau DF, Chen R, Wargo JJ, Rohan CA, Southern D, Zhang A, Loesch M, Weyerbacher J, Tholpady SS, Lewis DA, Kuhar M, Tsai KY, Castellanos AJ, Kemp MG, Markey M, Cates E, Williams AR, Knisely C, Bashir S, Gabbard R, Hoopes R, Travers JB. Randomized controlled trial of fractionated laser resurfacing on aged skin as prophylaxis against actinic neoplasia. J Clin Invest. 2021 Oct 1;131(19):e150972. doi: 10.1172/JCI150972. PMID 34428179
- [Derived] Chen R, Wargo JJ, Williams A, Cates E, Spandau DF, Knisely C, Travers JB. Single Ablative Fractional Resurfacing Laser Treatment For Forearm Actinic Keratoses: 6-Month Follow-Up Data From An Intrapatient Comparison Between Treated and Untreated Sites. Lasers Surg Med. 2020 Jan;52(1):84-87. doi: 10.1002/lsm.23175. Epub 2019 Nov 17. PMID 31736123

DOCUMENTS (1):
  • Informed Consent Form (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT03906253/ICF_000.pdf